CLINICAL TRIAL: NCT06110637
Title: Effects of Running Shoe Sole Hardness on Vibration and Neuromuscular Fatigue During a Half-marathon Run on a Treadmill
Acronym: FAT-VIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 21CH248; 2022-A00219-34 (Other: ANSM)
Record Dates: First submitted 2023-07-18; First posted 2023-10-31 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: Soft-tissue vibrations; Footwear; Endurance athletes; Running; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hard shoes runners (Experimental): Half-marathon runners with hard shoes preceded and followed by assessment of neuromuscular fatigue.
  Interventions: Other: "hard shoes" runners evaluation
- Soft shoes runners (Active Comparator): Half-marathon runners with soft shoes preceded and followed by assessment of neuromuscular fatigue.
  Interventions: Other: "Soft shoes" runners evaluation

INTERVENTIONS:
Other: "hard shoes" runners evaluation — The "hard shoes" runners get on the treadmill for 21 km at a speed corresponding to 70 percent (%) of their the maximum aerobic speed (MAV) and are evaluated.
  Arms: Hard shoes runners
Other: "Soft shoes" runners evaluation — The "soft shoes" runners get on the treadmill for 21 km at a speed corresponding to 70 percent (%) of their the maximum aerobic speed (MAV) and are evaluated.
  Arms: Soft shoes runners

SUMMARY:
During running, each contact between the foot and the ground causes an impact. Ground reaction forces (GRF) are considered as an input into the musculoskeletal system. It involves a sudden deceleration in the lower limb packages (including muscles) which generates Soft-Tissue Vibrations (STV). The body is able to attenuate Soft-Tissue Vibrations (STV) but this capability decreases with fatigue. STV could be minimize by improving shoe midsole hardness.

DETAILED DESCRIPTION:
Only 4 studies have studied Soft-Tissue Vibrations (STV) with a distance not exceeding 10 km and without evaluating the potential influence of the shoe. Thus, the effects of shoe midsole hardness on Soft-Tissue Vibrations (STV) and neuromuscular fatigue at the end of an intense and/or long run remains unknown.

The purpose is to compare two shoes whose only midsole hardness differs during a half-marathon on Soft-Tissue Vibrations (STV), neuromuscular fatigue and running kinetics.

Maybe the shoe ensuring a better STV damping of the medial gastrocnemius muscle would reduce neuromuscular fatigue and improve comfort.

ELIGIBILITY:
Inclusion Criteria:

* Endurance runners doing a long run of at least 20 km once a week.
* Affiliated or beneficiaries of a social security plan.
* Have freely given their written consent.
* Not participating in a competition during the study period.
* Shoe size 37 to 46

Exclusion Criteria:

* Any subject who has been injured in the 3 months preceding the protocol
* Any subject with chronic joint pathologies (e.g., repeated sprains, patellar or ligament problems) or cardiac pathologies.
* Any subject with chronic or central neurological pathologies
* Any subject participating at the same time in another medical interventional experiment
* Any subject who has taken corticosteroids within 3 months (inhalation, infiltration or history of prolonged corticosteroid therapy).
* Any subject deprived of liberty or under legal protection (guardianship, curatorship, safeguard of justice, family habilitation).
* Any subject declaring to have taken products prohibited by the World Anti-Doping Agency

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Change of the damping coefficient (in percent %). | From the beginning to the end of the 21 km race.
  The main evaluation criterion will be the relative variation (in percent %) of the damping coefficient (in /s) of the medial gastrocnemius muscle measured with an accelerometer, at the beginning (the first five minutes) and at the end (the last five minutes) of 21 km at a speed corresponding to 70% of the maximum aerobic speed (MAS) on a treadmill, carried out by experienced amateurs during two shoe conditions: soft and firm sole.

SECONDARY OUTCOMES:
Temporal evolution of vibrations measurements. | Kilometers : 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st
  The relative variation (in percent %) of the damping coefficient (in /s) of the medial gastrocnemius muscle will be measured with an accelerometer every 3 km at a speed corresponding to 70% of the maximum aerobic speed (MAS) on a treadmill, carried out by confirmed amateurs during the two shoe conditions.
  For this outcome, it is not possible to use an unit of time, because the time of the measurements are define only by the distance covered by the subject.
Evaluation of improved vibration damping on neuromuscular fatigue : isometric force | From the beginning to the end of the 21 km race.
  The relative change (in percent %) in the maximum isometric force (in Newton) of the ankle plantar flexors before and after the 21 km
Evaluation of improved vibration damping on neuromuscular fatigue : jerk amplitude. | From the beginning to the end of the 21 km race.
  The relative change (in percent %) in jerk amplitudes measured by electrically evoked force (in Newton) after isometric contraction of the plantar flexors of the ankle, before and after the 21 km.
Evaluation of improved vibration damping on neuromuscular fatigue : level of voluntary activation. | From the beginning to the end of the 21 km race.
  The relative change (percent %) in the maximum level of voluntary activation (percent %) measured in isometric mode of the plantar flexors of the ankle before and after the 21 km
Evaluation of improved vibration damping on neuromuscular fatigue : plantar flexors. | From the beginning to the end of the 21 km race.
  The relative change (in percent %) in the maximum isometric force (in Newton) of the plantar flexors of the toes before and after the 21 km.
Biomechanical parameters measurement : Ground reaction forces (Newton) | Kilometers : 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st.
  Ground reaction forces (in Newton, measured by treadmill force platforms).
  For this outcome, it is not possible to use an unit of time, because the time of the measurements are define only by the distance covered by the subject.
Biomechanical parameters measurement : Spatio-temporal parameters (second) | Kilometers : 1st, 3rd, 6th, 9th, 12th, 15th, 18th, 21st.
  Spatio-temporal parameters: contact time (CT) and flight time (TV)
  For this outcome, it is not possible to use an unit of time, because the time of the measurements are define only by the distance covered by the subject.
Temporal evolution of the energy cost measurement | From the beginning to the end of the 21 km race.
  This will be the relative variation (in percent %) of the energy cost (in J/kg/m), measured continuously thanks to a portable gas exchange measurement system (ergo spirometer Metamax 3B®, Cortex Medical, Leipzig, Germany), at a speed corresponding to 70% of the maximum aerobic speed (MAS) on a treadmill, carried out by experienced amateurs during the two shoe conditions.

CONTACTS AND LOCATIONS:
Overall Officials: LEONARD FEASSON, MDPHD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No